CLINICAL TRIAL: NCT05060796
Title: A Single-arm, Open-label, Phase I Study to Evaluate the Safety and Efficacy of CXCR5 Modified EGFR Chimeric Antigen Receptor Autologous T Cells in EGFR-positive Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Study of CXCR5 Modified EGFR Targeted CAR-T Cells for Advanced NSCLC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZBGCART-014
Record Dates: First submitted 2021-09-19; First posted 2021-09-29 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EGFR CAR-T (Experimental): Group: 3 dose levels
  Interventions: Biological: CXCR5 modified EGFR Chimeric Antigen Receptor Autologous T cells

INTERVENTIONS:
Biological: CXCR5 modified EGFR Chimeric Antigen Receptor Autologous T cells — The first dose group: 0.5 × 10^6/kg CAR positive T cells; The second dose group: 1.58 × 10^6/ kg CAR positive T cells; The third dose group: 5 × 10^6/kg CAR positive T cells. The above dose allows a 20 % error; For subjects with body weight greater than 60 kg, the number of cells can only be calculated according to 60 kg of body weight.

SUMMARY:
This study is a single arm, open-label, intravenous infusion of Anti- Epidermal growth factor receptor (EGFR) Chimeric Antigen Receptor (CAR) T cells modified by C-X-C Chemokine receptor type 5 (CXCR 5) in patients with advanced adult non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
In this study, the dose(number of cells by body weight) and time of infusion should be recorded in detail according to the dosage of slope climbing and single infusion. The safety of chimeric antigen receptor T(CAR-T) cells treatment was evaluated by observing the adverse events after cell therapy. The effectiveness of CAR-T treatment was initially assessed compared with the results of the patient's own previous standard treatment plan. Blood was collected before and within 12 months after infusion to detect the number and activity of CAR-T cells and evaluate the pharmacokinetic characteristics of CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects or legal guardians must sign the informed consent form approved by the ethics committee in writing before starting any screening procedure;
2. 18 Years to 75 Years, Histologically or cytologically confirmed Routine treatment of patients with advanced non-small cell lung cancer(Including TKI treatment failure patients);
3. After the signature of the informed consent and prior to the collection of a single nuclear cell, the immuno- histochemical test must determine that the expression of EGFR in the tumor site of the patient reaches the positive standard and the score is 2 + or more;
4. Pathological results suggest that CXCL13 factor positive rate ≥ 10 %;
5. According to RECIST 1.1. The patient has at least one tumor lesion that can be measured (Results available within one month prior to screening period);
6. Expected survival time ≥ 12 weeks;
7. The Eastern oncology group strength status score (ECOG) was 0-1;
8. Patients must have evidence of adequate hepatic and renal function as evidenced by the following laboratory parameters: Serum creatinine≤ 1.6 mg/ml or the creatinine clearance ≥ 40 ml/min/1.73m. Total bilirubin < 1.5 times upper limits of normal;
9. The hemodynamics determined by echocardiography or multichannel radionuclide angiography(MUGA) are stable and the left ventricular ejection fraction (LVEF)≥50%;
10. Have sufficient bone marrow reserves (subjects can meet this requirement through blood transfusion), defined as: The number of white blood cells should not be less than 2 × 10^9/L;Platelet≥100 x 10^9/L; Hemoglobin ≥100 g/L;
11. If the patient uses the following drugs, the following conditions must be met:

    Glucocorticoid: The therapeutic dose of glucocorticoid must be stopped 2 weeks before the EGFR CAR-T infusion. However, the following physiological replacement doses of glucocorticoids are allowed: 12 mg/m2 / dihydrogenated cortisone or equivalent; Immunosuppressive drugs: any immunosuppressive drugs must be stopped before they are selected for 4 weeks; Stop using granulocyte colony factor a week before plasmaphoresis.
12. Women of childbearing age and all male subjects must agree to use effective contraceptive methods for at least 52 weeks after EGFR CAR-T infusion, and until two consecutive PCR tests show that CAR-T cells are no longer present in the body.

Exclusion Criteria:

1. Patients who have previously received any gene therapy product treatment, including CAR-T treatment;
2. Patients with uncontrolled hypertension (> 160/95), unstable coronary artery disease confirmed by uncontrolled arrhythmias, unstable angina, decompensated congestive heart failure(>New York Heart Association Class II) or myocardial infarction within 6 months before cell infusion;
3. Patients with severe liver and kidney dysfunction or consciousness disorders;
4. Patients who had undergone antitumor chemotherapy other than lymphocyte clearance chemotherapy within 14 days before the EGFR CAR-T infusion;
5. Screening of patients who had received other research drugs within 30 days before infusion;
6. Patients undergoing radiotherapy and TKI treatment within 2 weeks before infusion ;
7. Patients with active hepatitis B: HBVDNA >1000 cps/ml;
8. Patients with HIV antibody, hepatitis C antibody, syphilis spirocyte positive；
9. Patients with The sputum smear and tuberculosis infection T cell test positive;
10. Patients with Interstitial lung disease or pneumonia;
11. Patients with acute life-threatening bacteria, viruses or fungal infections that have not yet been controlled(for example, before transfusion ≤ 72 hours of blood culture positive);
12. Patients with central nervous system metastasis (after cerebral metastasis treatment is stable for more than 4 weeks and patients with asymptomatic brain metastasis do not need treatment), pericardial metastasis accompanied by a large amount of pericardial effusion;
13. Patients with a previous or concurrent second tumor, with the following exceptions:

    Adequate treatment of basal or squamous cell carcinoma(adequate wound healing prior to entry into the study);In situ cancer of the cervix or breast cancer with no signs of recurrence at least three years prior to the study following curable treatment; The primary malignant tumor has been completely removed and has been completely relieved for 5 years.
14. Pregnant or lactating women;
15. Patients with history of T cell tumors or present with the disease.
16. Having autoimmune or inflammatory disorders of active nerves (such as Guillian-Barre syndrome, amyotrophic lateral sclerosis);
17. The researchers believe that other circumstances such as compliance should not be involved in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2034-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | In CAR-T cells infusion, up to 52 weeks.
  The type, frequency, severity, and duration of adverse events as a result of EGFR CAR T cells infusion will be summarized.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | In CAR-T cells infusion, up to 52 weeks.
  Per Response Evaluation Criteria in Solid Tumours (RECIST 1.1) assessed by MRI or CT. ORR is the percentage of patients at Complete Response (CR) or Partial Response (PR) (according to independent review), prior to progression or further anti-cancer therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PHD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No